CLINICAL TRIAL: NCT02641366
Title: Noninvasive Electromagnetic Tracking of Upper Extremity Motion Kinetics for Patients With Severe Tremor Disorders
Brief Title: Electromagnetic Tracking to Measure Tremor
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500964
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Tremor
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tremor kinetics after DBS: This group have already undergone Deep Brain Stimulation (DBS) placement and will have measurements of tremor kinetics by using the electromagnetic tracking. The electromagnetic sensors will be placed on the arm and hand while the routine outpatient neurologic examinations are being performed. The testing will be performed with the DBS system in both the on and off settings.
  Interventions: Device: Electromagnetic tracking; Procedure: Tremor kinetics after DBS
- Tremor kinetics before and after DBS: This group will have measurements of tremor kinetics by using electromagnetic tracking prior to being scheduled to undergo Deep Brain Stimulation (DBS) placement. A total of two testing sessions will be performed: the first session will be performed during the routine preoperative visit, the second session will be performed during the routine postoperative DBS programming visit in both the DBS on and the DBS off settings.
  Interventions: Device: Electromagnetic tracking; Procedure: Tremor kinetics before and after DBS

INTERVENTIONS:
Device: Electromagnetic tracking — The electromagnetic tracking system will precisely measure the position of a patient's upper extremity in space during routine neurologic examination.
Procedure: Tremor kinetics after DBS — We will fit the patient with the electromagnetic sensors and then perform routine outpatient neurologic examinations with their DBS system in both the DBS on and the DBS off settings.
  Groups: Tremor kinetics after DBS
Procedure: Tremor kinetics before and after DBS — We will perform two testing sessions: the first session will be performed during a routine preoperative visit, the second session will be performed during a routine postoperative DBS programming visit in both the DBS on and the DBS off settings.
  Groups: Tremor kinetics before and after DBS

SUMMARY:
Deep Brain Stimulation (DBS) is an effective treatment option for individuals with debilitating tremors that do not respond to medical therapy. However, severe tremors, particularly those that develop after central nervous system insult or from multiple sclerosis, can be comprised of several underlying components that represent dysfunction within distinct brain circuits. Some of these dysfunctional brain circuits can be successfully treated with DBS while others respond poorly DBS therapy. For severe tremors, it can be very difficult to discriminate between the underlying components of a patient movement disorder and is exclusively dependent upon clinical expertise. Even with extensive clinical experience, it is difficult to reliably predict the results of DBS therapy for patients suffering from severe, debilitating tremor. In an attempt to gain more knowledge, an electromagnetic tracking system will be used which can precisely measure the position of a patient's upper extremity in space during routine neurologic examination. The goal is to use this tool to quantitatively identify various components of severe tremor, which can be discriminated based on oscillatory frequency and regularity of tremor amplitude. The purpose of this research study is to better understand the nature of complex, severe tremors by carefully measuring movement of the upper extremities with sensors during simple tasks. The goal is to break down complicated tremors into their components and then determine which components will respond to deep brain stimulation.

DETAILED DESCRIPTION:
As a participant in the research study small sensors that are connected to wires will be affixed to points on your hand, wrist, elbow and/or shoulder. These sensors are painless and otherwise noninvasive. They will be used to measure the precise location of the hand and arm in space during the neurologic examination. This exam will test the tremors during short, simple tasks using the hand and arm. This information will be stored along with your name and medical record number for analysis after your testing is complete.

The sensors that are used to measure movements are connected to thin, flexible wires that will be attached with adhesive tape. The motion sensors use a magnet that produces a weak electromagnetic field. This electromagnetic field poses no direct harm, but could potentially interfere with medical devices such as cardiac pacemakers or deep brain stimulators if placed very close to the electromagnetic emitter.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Individuals who have undergone or are scheduled to undergo Deep Brain Stimulation (DBS) placement

Exclusion Criteria:

* Individuals who have not had or are not scheduled for Deep Brain Stimulation (DBS) placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 years old who have undergone deep brain stimulator implantation or are being considered for deep brain stimulation for severe, intractable tremor.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Power spectrum peaks | 1 day
  We will perform power spectrum analysis of raw movement data (X, Y, Z coordinates at each time point). Spectral analysis will be used to differentiate multiple underlying components of a patient's tremor that occur at different frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Oliveria, MD,PhD, Principal Investigator — University of Florida
Locations (1):
- Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No